CLINICAL TRIAL: NCT06526936
Title: The Effect of Foot Care Training Given to Diabetic Hemodialysis Patients on Foot
Brief Title: The Effect of Foot Care Training Given to Diabetic Hemodialysis Patients on Foot Care Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Ülkü YILMAZ, PHD, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: US2024
Record Dates: First submitted 2024-07-17; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Foot
Keywords: Diabetic Foot; Diabetes; Foot Care; Hemodialysis
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Training will be provided on diabetic foot care.
  Interventions: Behavioral: Education
- Control group (No Intervention): Since it is a control group, no application will be made.

INTERVENTIONS:
Behavioral: Education — Information about diabetic foot care
  Arms: Experimental group

SUMMARY:
Diabetic foot causes hospitalization, amputation and serious health problems in individuals. This situation also leads to loss of productivity of the individual, negatively. diabetic foot can be reduced by 85% with good foot care, education and a multidisciplinary team approach. Diabetes is observed in the majority of hemodialysis patients. Foot care becomes even more important if you have more than one chronic disease. The aim of this study is; To determine the effect of "Diabetic foot care training" given to diabetic hemodialysis patients on foot care behavior. The study was planned as a randomized controlled experimental study. It was planned for diabetic hemodialysis patients who were treated in a dialysis center with a study permit.

DETAILED DESCRIPTION:
Diabetic foot causes hospitalization, amputation and serious health problems in individuals. This situation also leads to loss of productivity of the individual, negatively affecting mental health and quality of life; It creates a serious economic burden on the family and healthcare system. However, it is stated that the development of diabetic foot can be reduced by 85% with good foot care, education and a multidisciplinary team approach. Diabetes is observed in the majority of hemodialysis patients. Foot care becomes even more important if you have more than one chronic disease. The aim of this study is; To determine the effect of "Diabetic foot care training" given to diabetic hemodialysis patients on foot care behavior. The study was planned as a randomized controlled experimental study. It was planned for diabetic hemodialysis patients who were treated in a dialysis center with a study permit. The population of the research consists of 64 diabetic hemodialysis patients. The sample consists of individuals who agreed to participate in the study. Number, percentage, mean and standard deviation will be used as descriptive statistical methods in the evaluation of the data. A normal distribution test will be applied to determine whether the research variables have a normal distribution. In case the research variables do not show normal distribution (p<0.05). In the analysis of variables for which the normality assumption is not met, non-parametric analysis methods Mann Whitney U (for comparisons of two groups) and Kruskal Wallis (for comparisons of three or more groups) will be used. Spearman correlation analysis will be performed to determine the relationship between the continuous variables of the research.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Having a diagnosis of diabetes
* Volunteering to participate in the study
* Good communication skills and the patient's ability to receive training himself

Exclusion Criteria:

* Not willing to participate in conflict

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-06-13 (Estimated); Study Completion 2025-06-13 (Estimated)

PRIMARY OUTCOMES:
Developing foot care behavior | Trainings are 15-20 minutes, once a week. 8 weeks in total will be given as.
  Providing training with diabetic foot care guidance As data collection forms in the research; The Participant Information Form prepared by the researcher and the Foot Care Behavior Scale (FBS) will be used.
  The lowest score that can be obtained on the scale is 15; The highest score is 75. The Cronbach alpha value of the scale was found to have high reliability as 0.83.

CONTACTS AND LOCATIONS:
Overall Officials: ULKU YILMAZ, Principal Investigator — Istanbul Beykent University
Locations (1):
- Idm Dialysis Center, Beylikduzu, Cumhuriyet Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No